CLINICAL TRIAL: NCT04465747
Title: Egyptian Liver Library: Rebuilding the Pyramid of Liver Disease Evidence in Egypt
Acronym: ELL
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Alboraie, Postgraduate clinical researcher, Al-Azhar University
Other Study IDs: MB-2
Record Dates: First submitted 2016-01-30; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Publications — Reviewing published evidence

SUMMARY:
A lot of publications about liver disease are available worldwide. Egypt is one of the countries having a large number of publications in hepatology. There are defects in reviewing this evidence and making use of it. Addressing the areas of weakness in liver research in Egypt is challenging to researchers and clinicians. Creating a library for liver disease evidence in Egypt can solve this problem and lead future research in hepatology in Egypt.

DETAILED DESCRIPTION:
Egypt is considered one of the countries with large liver disease burden in the world being endemic with bilharziasis and hepatitis C for decades. Limitations in health care resource further augment the magnitude of the problem allowing the development of disease specific complications in absence of effective treatments over the past. With discovery of anti-schistosomal therapy and implementation of the national program for eliminating bilharziasis; bilharzial liver disease incidence regressed markedly. However; complications of bilharzial liver disease are still present. The situation has been repeated with hepatitis C which is still a major health problem in Egypt regardless of the availability of highly effective interferon free antiviral regimens. This is mainly due to the large number of infected patients (estimated to be more than 6 million) [1], re-infection and presence of complications that needs further management. The need for addressing these major health problems in Egypt provoked a lot of research in the field of hepatology. Egyptian and non-Egyptian researchers have published a lot of scientific reports about liver diseases in Egypt. Since the ancient age of the pharaohs there were written evidence about liver disease in Egypt. It was reported in the Ebres Papyrus (around 2600 BC) that hardness of the liver occurs secondary to excess alcohol ingestion [2]. This was one of the oldest documented detailed medical literatures in the history of mankind. In the recent age there were a lot reports from Egypt about bilharziasis and other parasitic infestations as the one published by Cobbold in 1982 about injurious parasites in Egypt [3]. Further enormous amount of publications has been released afterwards. Reviewing this evidence and creating an indexed data base for it could be of value for the national and international hepatology platforms. I aim with other colleagues at reviewing all published evidence in the field of hepatology from Egypt up to January 2016 and classifying it by different key words to build a data base of liver disease evidence in Egypt. This data base will be continuously updated by published data after January 1st 2016 and will be the reference for researchers from Egypt and rest of the world. The data base will invite all authors from Egypt to provide their raw data of published articles to be available for further analyses by other researchers. Moreover the data base work team will start a series of systematic reviews and meta analyses for the available relevant data aiming at addressing the areas of strength and areas of weakness in liver disease research in Egypt making further recommendations to the research authorities about what is missing and how it is better to be addressed in their future research calls. This pilot research work can be reproduced elsewhere by other researchers in their own countries making use of their published data and advising their local research authorities to fill up the gaps in liver research in their own countries. Hopefully in the near future we will have these groups working together in a network driving liver research globally.

ELIGIBILITY:
Inclusion Criteria:

* Published articles about liver disease up to January 2016

Exclusion Criteria:

* Anything else

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Published articles about liver disease up to January 2016
Sampling Method: Non-Probability Sample
Enrollment: 5068 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Review of all published articles about liver disease in Egypt till April 2017 | 1 year
  Indexing articles according to types of liver disease

SECONDARY OUTCOMES:
Identifying missing diseases in hepatology research in Egypt | 1 year
  Identifying missing diseases in hepatology research in Egypt

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Alboraie, M.D., MRCP, Principal Investigator — Al-Azhay University, Cairo, Egypt
Locations (1):
- Al-Azhar Uinversity, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruggmann, P., Berg, T., Øvrehus, A. L. H., Moreno, C., Brandão Mello, C. E., Roudot-Thoraval, F., Marinho, R. T., Sherman, M., Ryder, S. D., Sperl, J., Akarca, U., Balık, İ., Bihl, F., Bilodeau, M., Blasco, A. J., Buti, M., Calinas, F., Calleja, J. L., Cheinquer, H., Christensen, P. B., Clausen, M., Coelho, H. S. M., Cornberg, M., Cramp, M. E., Dore, G. J., Doss, W., Duberg, A. S., El-Sayed, M. H., Ergör, G., Esmat, G., Estes, C., Falconer, K., Félix, J., Ferraz, M. L. G., Ferreira, P. R., Frankova, S., García-Samaniego, J., Gerstoft, J., Giria, J. A., Gonçales, F. L., Gower, E., Gschwantler, M., Guimarães Pessôa, M., Hézode, C., Hofer, H., Husa, P., Idilman, R., Kåberg, M., Kaita, K. D. E., Kautz, A., Kaymakoglu, S., Krajden, M., Krarup, H., Laleman, W., Lavanchy, D., Lázaro, P., Marotta, P., Mauss, S., Mendes Correa, M. C., Müllhaupt, B., Myers, R. P., Negro, F., Nemecek, V., Örmeci, N., Parkes, J., Peltekian, K. M., Ramji, A., Razavi, H., Reis, N., Roberts, S. K., Rosenberg, W. M., Sarmento-Castro, R., Sarrazin, C., Semela, D., Shiha, G. E., Sievert, W., Stärkel, P., Stauber, R. E., Thompson, A. J., Urbanek, P., van Thiel, I., Van Vlierberghe, H., Vandijck, D., Vogel, W., Waked, I., Wedemeyer, H., Weis, N., Wiegand, J., Yosry, A., Zekry, A., Van Damme, P., Aleman, S. and Hindman, S. J. (2014), Historical epidemiology of hepatitis C virus (HCV) in selected countries. Journal of Viral Hepatitis, 21: 5-33. doi: 10.1111/jvh.12247
- [Result] Starr SP, Raines D. Cirrhosis: diagnosis, management, and prevention. Am Fam Physician. 2011 Dec 15;84(12):1353-9. PMID 22230269
- [Result] Cobbold TS. Remarks on Injurious Parasites of Egypt in Relation to Water-Drinking. Br Med J. 1882 Sep 16;2(1133):503-4. doi: 10.1136/bmj.2.1133.503. No abstract available. PMID 20750313